CLINICAL TRIAL: NCT07187349
Title: A Scalable Intervention for Stress Management Real World Assessment
Brief Title: Real World Assessment of Resistance Breathing Device
Status: Not yet recruiting | Type: Observational
Sponsor: Livotion, LLC (Industry)
Collaborators: Purdue University (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB-2025-13; 1R41AT012854-01 (NIH)
Record Dates: First submitted 2025-09-18; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Stress; Breathing Exercise; Stress Management
Keywords: Stress management; Resistance breathing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Undergraduate Exam Takers: College undergraduate students between the ages of 18-30 who will be involved in an academic examination period at Purdue University.

SUMMARY:
The purpose of this study is to examine the usability and effectiveness of a stress management device during an academic exam period and asks the following questions:

* To what extent is a resistance breathing device (AIRpen) utilized by participants during the study period?
* What impact does utilizing a resistance breathing device have on participant's well-being when used during a stressful academic period?
* To what extent is a diaphragmatic breathing device acceptable for use when utilized during a noted stress-inducing period such as academic examinations?

DETAILED DESCRIPTION:
This study aims to build upon prior work with a diaphragmatic breathing intervention, testing the acceptability and usability of a resistance breathing device for stress reduction (i.e., the AIRpen) amongst college students during the academic semester. Regulated breathing has been shown to be an accessible and effective form of stress reduction, with prior research identifying diaphragmatic breathing as a key form of stress reduction that can impart cognitive, emotional, and physical benefits. Accomplishing diaphragmatic breathing can be difficult however, as it is a skill which requires considerable practice and can be challenging to perform properly without assistance.

To address this, a number of eHealth and physical applications (e..g, inhalers, mediations apps, chest straps) have arisen which seek to assist individuals in regulating their breathing and facilitating diaphragmatic breathing. However, the suitability of such interventions varies greatly, and may not always be appropriate for different contexts. For college students especially, a group which experiences a wide range of stressors within the course of their studies, interventions such as eHealth mobile applications or inhalers may be cumbersome, contextually inappropriate, or potentially stigmatizing when utilized within their educational environment. To address this, the PI has developed the AIRpen, a simple, affordable, and multi-functional stress management and regulated breathing device which aims to blend into a student's environment and assist in achieving diaphragmatic breathing in a discreet and effective manner. With anecdotal and empirical evidence supporting the device as feasible and acceptable in real-world academic settings (Purdue IRB-2022-423), this study will build upon prior work and measure the acceptability and feasibility of the AIRpen, as well as it's effect on perceived stress and coping self-efficacy amongst college students. As the purpose of this study, which is being funded by the NIH, is to study use of the AIRpen amongst college aged individuals, college students are not a convenience sample but actually the target sample for the study.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old
* Be currently enrolled in a college or university
* Be able to read, speak, and comprehend English
* Be able and willing to complete a 2-week long study involving survey completion, training, and AIRpen utilization during an academic examination period

Exclusion Criteria:

- Individuals with a diagnosis of anxiety or stress that require professional support to cope with such clinical levels of stress or anxiety should not enroll in the study in place of professional assistance

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Undergradute students from Purdue University
Sampling Method: Non-Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2025-10-13 (Estimated); Primary Completion 2025-11-07 (Estimated); Study Completion 2025-11-07 (Estimated)

PRIMARY OUTCOMES:
Device Usability as Measured by a Modified Version of the System Usability Scale (SUS) | From study enrollment to the end of the study at 2 weeks.
  The System Usability Scale is a 10-item measure that address the usability and learnability of a system. The SUS has been modified to reflect the AIRpen intervention. Statements are ranked on a Likert scale for 1-5, with 1 indicating "Strongly Disagree" and 5 indicating "Strongly Agree". Raw scores are converted into a final score that ranges from 0-100, with a larger score indicating greater usability.
Device Acceptability as Measured by the Acceptability of Intervention Measure (AIM) | From study enrollment to the end of the study at 2 weeks.
  The AIM measure is designed to assess the acceptability of a intervention, and has been adapted in relation to the AIRpen. Participants rate statements related to their usage and experience of the AIRpen and AIRpen website, with ratings ranging from "Completely Disagree" (1), to "Completely Agree" (5). Higher scores indicate higher acceptability of the intervention.
Device Feasibility as Measured by the Feasibility of Intervention Measure (FIM) | From study enrollment until the end of the study at 2 weeks.
  The Feasibility of Intervention Measure (FIM) measures the feasibility of an intervention through a 5-point Likert scale, and has been adapted in relation to the AIRpen. Statements relate to the overall feasibility of the intervention, with 1 indicating "Completely disagree" while 5 indicates (Completely agree), with a higher score indicating greater feasibility.

SECONDARY OUTCOMES:
Problem-Focused Coping as Measured by the Coping Self-Efficacy Scale (CSES) | From study enrollment to the end of the study at 2 weeks
  The Coping Self-Efficacy Scale (CSES) measures an individual's degree of confidence that s/he can perform coping behaviors when faced with life challenges. The CSES consists of three subscales measuring Problem-focused Coping, Emotion-focused Coping, and Social Support Coping. The CSES is administered as a 26-item form, although for this study only the Problem-Focused Coping subscale is administered.
Perceived Stress as Measured by the Perceived Stress Scale (PSS_10) | From study enrollment to the end of the study at 2 weeks.
  The Perceived Stress Scale is a measure used to assess perceptions of recent stress. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.

IPD SHARING:
Plan to Share IPD: No